CLINICAL TRIAL: NCT04975022
Title: Research on Clinical Application of New Therapies for Diabetes and Its Complications and Related Translational Medicine Research
Brief Title: A Study Evaluating the Bioavailability of Oral Insulin (N11005)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 12013-P-01
Record Dates: First submitted 2021-07-21; First posted 2021-07-23 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: PK, PD, and Safety
MeSH Terms: interventions — Insulin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T group (Experimental)
  Interventions: Drug: N11005
- R group (Active Comparator)
  Interventions: Drug: Novolin R

INTERVENTIONS:
Drug: N11005 — oral insulin N11005, 300IU, p.o.
  Arms: T group
Drug: Novolin R — reference preparation Novolin R, 0.1 IU/Kg, i.h.
  Arms: R group

SUMMARY:
The objective of this study was to preliminarily verify whether the oral insulin N11005 is a prandial insulin by assessing the PK, PD, and safety profiles of N11005.

ELIGIBILITY:
Inclusion Criteria:

* 1) Volunteer to participate in the trial and sign an informed consent form; 2) 18-45 years old (including 18 and 45 years old) healthy male subjects (without heart, liver, kidney, digestive tract, neurological diseases, and metabolic abnormalities in the 4 weeks before screening; No abnormal clinically significant vital signs results, physical examination results, laboratory examination results and electrocardiogram examination results judged by the investigator at the time of screening); 3) BMI (body mass index): between 19-24 Kg/m2, including 19 and 24 Kg/m2; 4) Normal glucose tolerance (fasting plasma glucose [FPG] <6.1 mmol/L, and oral glucose tolerance test [OGTT] 2-hour postprandial blood glucose <7.8 mmol/L); 5) No family history of diabetes, obesity, etc.; 6) Insulin secretion function is normal (confirmed by insulin release test (IRT) judged by the investigator); 7) There is no planned parenthood during the study period, and it is agreed to use reliable contraceptive measures during the study period until 4 weeks after the last administration of the study drug; 8) Be able to communicate well with researchers and complete research in accordance with research regulations.

Exclusion Criteria:

* 1). Those who have serious systemic diseases, infectious diseases or mental disorders; 2). The results of human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody, syphilis test are positive; 3). Those who have used any prescription drugs, Chinese herbal medicines and/or over-the-counter drugs (except for subjects with occasional and restricted use of paracetamol) and health products (except routine vitamin supplements) within 2 weeks before screening; 4). Those who donated more than 400 mL of blood within 3 months before screening; 5). Severe smokers (25 or more cigarettes per day); 6). Alcoholics (drinking 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine), or those who have a positive alcohol breath test result; 7). Those who have a history of drug abuse or have a positive urine test for illegal drugs; 8). Those who are known or suspected to be allergic to insulin and/or its excipients; 9). Those who have participated in other clinical trials within 3 months before screening, or plan to participate in other clinical trials during the trial period or within 1 month after the end of the trial; 10). Those who have any food allergies or have special dietary requirements and cannot follow a unified diet; 11). Those who have undergone gastrointestinal surgery before screening, or have a history of gastric obstruction or impaired gastrointestinal motility; 12). Those who are using gastric mucosal protective agents during screening; 13). Those who are deemed unsuitable to participate in this trial after the researcher's evaluation;

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
Cmax | Pre-dose, 5,10,20,30,40,50,60,75,90,105,120,150,180,210,240,270,300, 330,360,420,480 minutes；
  the peak concentration
AUC 0-8 h | Pre-dose, 5,10,20,30,45,10,20,30,40,50,60,75,90,105,120,150,180,210,240,270,300, 330,360,420,480 minutes；
  the AUC for insulin from time zero to 8 hours
AUCGIR,0-8 h | Pre-dose, 0-8 hours
GIRmax | Pre-dose, 0-8 hours

SECONDARY OUTCOMES:
Tmax | Pre-dose, 5,10,20,30,40,50,60,75,90,105,120,150,180,210,240,270,300,330,360,420,480 minutes；
  time to Cmax
AUC 0-2 h | Pre-dose, 5,10,20,30,40,50,60,75,90,105,120 minutes
  the AUC for insulin from time zero to 2 hours
the elimination half-life (t1/2) of serum insulin | Pre-dose, 5,10,20,30,40,50,60,75,90,105,120,150,180,210,240,270,300, 330,360,420,480 minutes；
the AUC for insulin from time zero to 4 h | Pre-dose, 5,10,20,30,40,50,60,75,90,105,120,150,180,210,240 minutes
the AUC for insulin from time zero to infinite time | Pre-dose, 5,10,20,30,45,10,20,30,40,50,60,75,90,105,120,150,180,210,240,270,300, 330,360,420,480 minutes；
AUCGIR，0-2 h | Pre-dose, 0-2 hours
AUCGIR，0-4 h | Pre-dose, 0-4 hours
tGIRmax | Pre-dose, 0-8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, China

REFERENCES:
- [Derived] Pan Q, Wang X, Li W, Chen X, Zhuang Y, Zhou Q, Huang Y, Zhou Y, Lan L, Wang Z, Wang W, Hong J, Hao WH, Yang YT, Guo L. Pharmacokinetics, pharmacodynamics, and safety of prandial oral insulin (N11005) in healthy subjects. Front Endocrinol (Lausanne). 2023 Jul 26;14:1172327. doi: 10.3389/fendo.2023.1172327. eCollection 2023. PMID 37564986